CLINICAL TRIAL: NCT06808698
Title: A Study of the Intestinal Microbiome in Patients with Cirrhosis
Acronym: IIT_MicroB
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hye Won Lee, Professor, MD, Yonsei University
Other Study IDs: IIT_MicroB
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA 5ml, SST 5ml
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with cirrhosis: Patients with cirrhosis
  Interventions: Other: Determine the gut microbiome at baseline and 12 months.

INTERVENTIONS:
Other: Determine the gut microbiome at baseline and 12 months. — There is no separate treatment, surgery, or other intervention.

SUMMARY:
This study aims to establish a cohort for analyzing the gut microbiome of patients with liver cirrhosis and to identify factors that influence the prognosis of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 years or older:
2. Patients visiting the hospital with liver cirrhosis.
3. Patients diagnosed with liver cirrhosis who can understand the information provided to them or their representatives and have voluntarily given written consent to participate in this study

Exclusion Criteria:

1. Cases not meeting the inclusion criteria
2. Patients who refuse participation
3. Patients who have taken or been administered antibiotics within the past 2 weeks or are scheduled to take or receive antibiotics during the study period
4. Cases where the diagnosis is unclear
5. Cases with incomplete data or missing investigation items
6. Individuals deemed unsuitable by the principal investigator for other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting our hospital with liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of non-targeted complications according to changes in the gut microbiome | baseline, Month 12
  We observed changes in the gut microbiome of the subjects participating in the study at baseline and 12 months, and confirmed the incidence of non-target complications accordingly.

SECONDARY OUTCOMES:
Liver cancer incidence rate according to gut microbiome composition | Baseline, 12 Month
  We observed changes in the gut microbiome of the subjects participating in the study at baseline and 12 months, and confirmed the liver cancer incidence rate accordingly.

IPD SHARING:
Plan to Share IPD: Undecided